CLINICAL TRIAL: NCT04284774
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice)- Phase 2 Subprotocol of Tipifarnib in Patients With Tumors Harboring HRAS Genomic Alterations
Brief Title: Tipifarnib for the Treatment of Advanced Solid Tumors, Lymphoma, or Histiocytic Disorders With HRAS Gene Alterations, a Pediatric MATCH Treatment Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01015; NCI-2020-01015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621M (Other: Children's Oncology Group); APEC1621M (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Malignant Solid Neoplasm; Recurrent Adrenal Gland Pheochromocytoma; Recurrent Ectomesenchymoma; Recurrent Ependymoma; Recurrent Ewing Sarcoma; Recurrent Hepatoblastoma; Recurrent Kidney Wilms Tumor; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Glioma; Recurrent Medulloblastoma; Recurrent Melanoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Rhabdoid Tumor; Recurrent Rhabdoid Tumor of the Kidney; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Recurrent Thyroid Gland Carcinoma; Recurrent WHO Grade 2 Glioma; Refractory Adrenal Gland Pheochromocytoma; Refractory Ependymoma; Refractory Ewing Sarcoma; Refractory Hepatoblastoma; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Glioma; Refractory Medulloblastoma; Refractory Melanoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Rhabdoid Tumor; Refractory Rhabdoid Tumor of the Kidney; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Refractory Thyroid Gland Carcinoma; Refractory WHO Grade 2 Glioma
MeSH Terms: conditions — Pheochromocytoma; Ependymoma; Sarcoma, Ewing; Hepatoblastoma; Wilms Tumor; Histiocytosis, Langerhans-Cell; Glioma; Medulloblastoma; Melanoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Thyroid Neoplasms | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive tipifarnib tablets 350 mg/m^2/dose PO or via nasogastric or gastric tube BID (maximum 600 mg/dose BID) with food on days 1-7 and 15-21. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — Tipifarnib tablets
  Other Names: R115777; Zarnestra

SUMMARY:
This phase II pediatric MATCH trial studies how well tipifarnib works in treating patients with solid tumors that have recurred or spread to other places in the body (advanced), lymphoma, or histiocytic disorders, that have a genetic alteration in the gene HRAS. Tipifarnib may block the growth of cancer cells that have specific genetic changes in a gene called HRAS and may reduce tumor size.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with tipifarnib with advanced solid tumors (including central nervous system [CNS] tumors), lymphomas or histiocytic disorders that harbor activating genetic alterations in HRAS.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with tipifarnib with advanced solid tumors (including CNS tumors), lymphomas or histiocytic disorders that harbor activating genetic alterations in HRAS.

II. To obtain information about the tolerability of tipifarnib in children and adolescents with relapsed or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate other biomarkers as predictors of response to tipifarnib and specifically, whether tumors that harbor different missense mutations or variant allele frequency will demonstrate differential response to tipifarnib treatment.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive tipifarnib tablets 350 mg/m^2/dose orally (PO) or via nasogastric or gastric tube twice daily (BID) (maximum 600 mg/dose BID) with food on days 1-7 and 15-21. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC (NCT03155620) and must have been given a treatment assignment to MATCH to APEC1621M based on the presence of an actionable mutation as defined in APEC1621SC
* Patients must be >=12 months and =< 21 years of age at the time of study enrollment
* Patients must have a body surface area >= 0.29 m^2 at enrollment
* Patients must have radiographically measurable disease at the time of study enrollment. Patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG) positive (+) evaluable disease are eligible. Measurable disease in patients with CNS involvement is defined as any lesion that is at minimum 10 mm in one dimension on standard magnetic resonance imaging (MRI) or computed tomography (CT)

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebral spinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Karnofsky >= 50 for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation

    * Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radio-pharmaceutical therapy
  * Patients must not have received prior exposure to tipifarnib
* For patients with solid tumors without known bone marrow involvement (within 7 days prior to enrollment):

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* For patients with solid tumors without known bone marrow involvement (within 7 days prior to enrollment):

  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 (within 7 days prior to enrollment) or
* A serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * Age: Maximum serum creatinine (mg/dL)

    * 1 to < 2 years: male (0.6), female (0.6)
    * 2 to < 6 years: male (0.8), female (0.8)
    * 6 to < 10 years: male (1), female (1)
    * 10 to < 13 years: male (1.2), female (1.2)
    * 13 to < 16 years: male (1.5), female (1.4)
    * >= 16 years: male (1.7), female (1.4)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. (For the purpose of this study, the ULN for SGPT is 45 U/L.) (within 7 days prior to enrollment)
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment)
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) resulting from prior therapy must be =< grade 2
* Patients must be able to swallow intact tablets or crushed tablets mixed in water, orange juice, apple juice, tomato juice, ginger ale, applesauce, yogurt, protein shake, or a dietary supplement drink (such as Ensure). Percutaneous endoscopic gastrostomy (PEG)-tube or nasogastric tube administration is permitted
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective contraceptive methods for the duration of study treatment. Both female subjects and male subjects with female partners of child-bearing potential must agree to use a highly effective method of contraception for 2 weeks prior to protocol therapy, during, and at least 4 weeks after last dose of tipifarnib. In addition, since tipifarnib could induce toxicity of male reproductive organs and cause impairment of fertility, sperm cryopreservation should be recommended for male subjects wishing to preserve their fertility following tipifarnib treatment
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4/5 or UGT are not eligible. Strong inducers or inhibitors of CYP3A4/5 or UGT should be avoided from 14 days prior to the 1st dose of tipifarnib to the end of the study. In addition, patients receiving agents that are sensitive or narrow therapeutic range substrates of CYP3A4/5 are not eligible. Note: CYP3A4/5 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed
* Patients with known hypersensitivity to tipifarnib or any components of the tablet are not eligible
* Patients with hypersensitivity to imidazoles, such as clotrimazole, ketoconazole, miconazole and others in this drug class are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2027-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Pratilas, Principal Investigator — Children's Oncology Group
Locations (172):
- United States (171):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between 10Oct2020 and 31Mar2024, 7 subjects matched and 5 were included and treated with study drug. Subjects received a median of 2 cycles of study drug (range 1-4 cycles).
Period: Overall Study
Arm/Group | Treatment (Tipifarnib)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Progressive disease | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tipifarnib)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response + Partial Response) in Pediatric Patients Treated With Tipifarnib
Description: A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method. The revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to determine response and progression in this study, with specific criteria outlined for the different subtypes of tumors (e.g., 2-dimensional measurements for central nervous system (CNS) tumors.
Time Frame: Up to 2 years from study entry
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Tipifarnib)
Number analyzed (Participants) | 5
percentage of patients | 0 [0 to 0]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the 6-month PFS. PFS is defined as time from initiation of protocol treatment to disease progression, recurrence, death from any cause, or date of last contact
Time Frame: Up to 6 months from study entry
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or Higher Adverse Events
Description: Percentage of patients experiencing grade 3 or higher adverse events will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0
Time Frame: Up to 2 years from study entry
Reporting Status: Not Posted, anticipated posting 2026-03

4. Other Pre Specified Outcome: Biomarker Analysis
Description: Will evaluate other biomarkers as predictors of response to tipifarnib and whether tumors that harbor different missense mutations or fusions will demonstrate differential response to treatment.
Time Frame: Up to 7 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Profiling Changes in Tumor Genomics
Description: Will explore approaches to the profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid.
Time Frame: Baseline, prior to cycle 5, end of treatment, assessed up to 7 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment to 30 days after the end of treatment, up to 2 years.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Tipifarnib)
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tipifarnib) (N=5)
Disease progression (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Tipifarnib) (N=5)
Anemia (Blood and lymphatic system disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04284774/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04284774/ICF_001.pdf